CLINICAL TRIAL: NCT00693316
Title: Phase I Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study With Single Ascending Doses of ORM-12741
Brief Title: Safety and Tolerability Study With Single Ascending Doses of ORM-12741
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Jutta Hänninen, Clinical study manager, Orion corporation, Orion Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3098001
Record Dates: First submitted 2008-05-30; First posted 2008-06-09 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORM-12741 (Experimental)
  Interventions: Drug: ORM-12741
- Placebo (Placebo Comparator)
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — Alternating panel single dose escalation.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating doses of ORM-12741 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Good general health ascertained by detailed medical history and physical examinations
* Males between 18 and 45 years
* Body mass index (BMI) between 18-30 kg/m2
* Weight 55-90 kg

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease
* Any condition requiring regular concomitant treatment including herbal products or likely to need any concomitant treatment during the study
* Susceptibility to severe allergic reactions
* Regular consumption of more than 14 units of alcohol per week
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day
* Inability to refrain from using nicotine-containing products during the stay in the study centre
* Inability to refrain from consuming caffeine-containing beverages during the stay in the study centre
* Blood donation or loss of significant amount of blood within 3 months prior to the screening visit
* Abnormal finding in ECG, vital signs, laboratory tests or physical examination
* Participation in a drug study within 3 months prior to the start of this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety measures, i.e. assessing adverse events, vital signs, ECG, safety laboratory values | About 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | 5 days after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Déborah Metzger, MD, Principal Investigator — Forenap Pharma
Locations (1):
- Forenap Pharma, Rouffach, France